CLINICAL TRIAL: NCT02030132
Title: A Randomized Trial of Behavioral Economic Interventions to Improve Physical Activities: Framing vs. Forgiveness
Brief Title: Way to Be Active V (Framing vs. Forgiveness)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 819370
Record Dates: First submitted 2013-12-20; First posted 2014-01-08 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Sedentary Lifestyle
Keywords: Physical activity; Sedentary lifestyle; Pedometers; Walking; Financial Incentives; Behavioral Economics
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Feedback 50th Percentile (Active Comparator): At the end of each week, participants will be told (by email or text, based on the participant's preference) the team's average daily step count for the previous week based on all 7 days. They will also be told the average for the 50th percentile in their arm. If the team's average daily step count is ≥ 7000 steps, the team will be eligible for the weekly lottery.
  Interventions: Behavioral: Financial Incentive; Behavioral: Daily Feedback
- Feedback 75th Percentile (Experimental): At the end of each week, participants will be told (by email or text, based on the participant's preference) the team's average daily step count for the previous week based on all 7 days. They will also be told the average for the 75th percentile in their arm. If the team's average daily step count is ≥ 7000 steps, the team will be eligible for the weekly lottery.
  Interventions: Behavioral: Feedback compared to 75th percentile; Behavioral: Financial Incentive; Behavioral: Daily Feedback
- Feedback 50th Percentile + Forgiveness (Experimental): At the end of each week, participants will be told (by email or text, based on the participant's preference) the average team's average daily step count for the previous week based on the best 5 of 7 days. They will also be told the average for the 50th percentile in their arm. If the team's average daily step count (best 5 of 7 days) is ≥ 7000 steps, the team will be eligible for the weekly lottery.
  Interventions: Behavioral: Forgiveness; Behavioral: Financial Incentive; Behavioral: Daily Feedback
- Feedback 75th Percentile + Forgiveness (Experimental): At the end of each week, participants will be told (by email or text, based on the participant's preference) the team's average daily step count for the previous week based on the best 5 of 7 days. They will also be told the average for the 75th percentile in their arm. If the team's average daily step count (best 5 of 7 days) is ≥ 7000 steps, the team will be eligible for the weekly lottery.
  Interventions: Behavioral: Feedback compared to 75th percentile; Behavioral: Forgiveness; Behavioral: Financial Incentive; Behavioral: Daily Feedback

INTERVENTIONS:
Behavioral: Feedback compared to 75th percentile
  Arms: Feedback 75th Percentile; Feedback 75th Percentile + Forgiveness
Behavioral: Forgiveness
  Arms: Feedback 50th Percentile + Forgiveness; Feedback 75th Percentile + Forgiveness
Behavioral: Financial Incentive — For the first three months of the study, a weekly lottery will be held. Teams whose average daily step count for that week is ≥ 7000 will be eligible to collect their lottery winnings. Teams whose average daily step count is less than 7000 will receive messages about how much they would have won had the team met its goal.
Behavioral: Daily Feedback — Participants will be given daily feedback on whether or not they walked 7000 steps or more the day before.

SUMMARY:
Employers are increasingly looking for opportunities to motivate sedentary employees to become more physically active. Workplace walking programs have had mixed success and typically show most improvement among participants that are already fairly active at a baseline. The goal of this study is to determine whether a financial incentive program can motivate sedentary employees to increase the number of steps they walk per day to meet a minimum threshold.

The primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. Outcomes will be assessed each week for 3 months using incentives followed by 3 months of follow-up without incentives. Secondary outcomes will include the average steps walked per day.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18.
* Participant will need an iPhone or Android smartphone to be able to use the Moves App for tracking steps

Exclusion Criteria:

* Pregnant or lactating
* Participating in another physical activity study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Proportion of days an individual walks 7000 steps or more | End of study - 6 months after enrollment
  The primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. Outcomes will be assessed each week for 3 months using incentives followed by 3 months of follow-up without incentives.

SECONDARY OUTCOMES:
Average number of steps per day and week | End of study- 6 months after enrollment
  Secondary outcomes include average number of steps per day and week during the intervention (first 3 months) and follow-up (second 3 months) periods.

OTHER OUTCOMES:
Change in physical activity | End of study- 6 months after enrollment
  Changes in physical activity as determined by validated surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; Mitesh Patel, MD, MBA, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States